CLINICAL TRIAL: NCT02195050
Title: Hypertriglyceridaemia: Therapeutic Targets, Genetic Causes, and Associated Neuropathy
Brief Title: Abnormal Lipids - Causes and Effects
Status: Recruiting | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: APOB2012; R03301 (Other: Manchester University NHS Foundation Trust)
Record Dates: First submitted 2014-07-10; First posted 2014-07-21 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Hypertriglyceridaemia
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum & plasma samples will be stored for further studies.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Therapeutic target arm: Statin treated patients with and without raised triglycerides who do not have diabetes or dysglycemia. Statin treated patients with type 2 diabetes.Statin treated patients with CKD stages 4 and 5 (eGFR ≤30mL/min).
- Nerve function arm: Patients with severe hypertriglyceridaemia (fasting TG > 5.5mmol/l.) are recruited for nerve function assessment and corneal confocal microscopy.
- Genetic screening arm: For LAL deficiency screening, patients will be recruited over a 5 year period with a documented triglyceride level of more than 10 mmol/l at any time, low HDLC, raised ALT, combined hyperlipidaemia, or non-alcoholic fatty liver disease. Patients recruited from Manchester will be offered additional genetic testing for familial hypercholesterolaemia.

SUMMARY:
1. At target LDL-C levels, apoB100 concentrations will be higher than recommended levels in the following populations:

   1. Tertiary centre lipid clinic patients with raised TG treated with statins.
   2. Patients with type 2 diabetes treated with statins.
   3. Patients with Chronic Kidney disease (CKD) stages 4 and 5 treated with statins.
2. Despite achieving LDL-C and non-HDL-C targets, a significant number of statin-treated patients have residual cardiovascular risk related to raised hsCRP. The relationship between hsCRP and Lp-PLA2 (markers of inflammation) and LDL particle number measured by apoB100 is stronger than that of measured and calculated LDL and non-HDL. In statin treated patients there will be higher levels of hs-CRP and Lp-PLA2 in patients achieving LDL targets but not apo B targets.
3. We hypothesise that non-diabetic patients with severe hypertriglyceridaemia (fasting serum triglyceride >5.5 mmol/l) have evidence of greater nerve damage compared with matched controls.
4. LAL deficiency is underdiagnosed in patients with severe hypertriglyceridaemia, low HDL-C, hyperlipidaemias, non alcoholic fatty liver disease and idiopathic high liver enzymes.

DETAILED DESCRIPTION:
Fats are present in the body in the form of lipid particles containing cholesterol and triglycerides. Lipid particles can deposit in blood vessels, forming atheromas, blocking blood vessels and leading to heart attacks and strokes. These harmful particles are termed 'atherogenic' particles. Low density lipoprotein (LDL) is the major atherogenic particle. Each atherogenic particle has a protein associated with it called apolipoprotein B (apoB). Cholesterol, triglycerides, and apoB levels can be measured in the laboratory. In this study we focus on patients with raised levels of triglycerides (hypertriglyceridaemia).

We will recruit patients with hypertriglyceridaemia to look at (1) therapeutic targets, (2) genetic causes, and (3) associated neuropathy in these patients.

1. Therapeutic target arm:

   LDL-cholesterol (LDL-C) is the primary target for lipid-lowering drugs. A drug (commonly a statin) is effective when it lowers LDL-C. Patients with diabetes, chronic kidney disease and hypertriglyceridaemia on statins may have normal levels of LDL-C; but because the size of LDL particles in these patients is smaller, they may in fact have raised levels of apoB and therefore remain at cardiovascular risk. Thus, measurement of apoB may be a better target for treatment because it measures 'atherogenic' particle numbers. Since atheromatous disease is an inflammatory disease, we will also investigate if residual risk may be correlated with inflammatory markers, such as hsCRP and Lp-PLA2.
2. Hypertriglyceridaemia and nerve function arm:

   We aim to demonstrate that severe hypertriglyceridaemia is associated with more significant nerve damage.
3. Genetic screening arm:

Several genetic mutations have been identified to cause hypertriglyceridaemia. Deficiency of the enzyme lysosomal acid lipase (LAL) results in Cholesterol Ester Storage Disease (CESD) and hypercholesterolaemia, hypertriglyceridaemia, and abnormal lipid deposition in organs. We wish to identify genetic mutations associated with severe hypertriglyceridemia and the prevalence of LAL deficiency in patients attending our tertiary referral centre.

ELIGIBILITY:
Inclusion Criteria:

* Therapeutic target arm

  * Statin treated patients with and without hypertriglyceridemia.
  * Statin treated patients with type 2 diabetes.
  * Statin treated patients with CKD stages 4 and 5.
* Nerve function arm

  •Patients known to have severe hypertriglyceridaemia (defined as triglyceride >5.5 mmol/l) but not known to have diabetes and matched controls.
* Genetic screening arm

  * Patients with a documented triglyceride level of more than 10 mmol/l at any time.
  * Criteria for screening for FH and LAL deficiency include non-obese patients (BMI <30) with low HDL-C (<1.0 mmol/l male and <1.3 mmol female), high triglycerides >1.7 mmol/l, high total cholesterol >6.2 or LDL cholesterol >4.7 mmol/l; patients with raised liver alanine aminotransferase (ALT) (1.5 x above ULN) but no metabolic or viral disease or alcohol excess and patients diagnosed with NAFLD with or without hyperlipidaemia.

Exclusion Criteria:

* Pregnant and/or breast-feeding women.
* Significant liver impairment.
* Patients known to have active malignant disease.
* Patients treated with medications that could affect lipoprotein metabolism significantly (like atypical antipsychotics, chemotherapy).
* Untreated hypothyroid and hyperthyroidism (if treated and TFT normal could be recruited).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are recruited from secondary and tertiary care hospital clinics.
Sampling Method: Non-Probability Sample
Enrollment: 1396 (Estimated)
Dates: Start 2014-01-23 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of ApoB in specified patient populations to gauge cardiovascular risk. | 1 day.
  Residual risk due to the presence of sd-LDL and reflected in a discrepancy between apoB and cholesterol indices is correlated with hs-CRP.

CONTACTS AND LOCATIONS:
Overall Officials: Handrean Soran, MD FRCP, Principal Investigator — Manchester University NHS Foundation Trust
Locations (1):
- Cardiovascular Trials Unit, Manchester, United Kingdom